CLINICAL TRIAL: NCT04279171
Title: Incidence of Near-death Experiences Among Patients Who Survived a Critical Illness
Brief Title: Near-death Experience in ICU Survivors
Status: Completed | Type: Observational
Sponsor: University of Liege (Other)
Responsible Party: Principal Investigator, Anne-Françoise Rousseau, Head of Clinic, Intensive Care Dpt, University of Liege
Other Study IDs: EMISI
Record Dates: First submitted 2020-02-19; First posted 2020-02-21 (Actual); Last update posted 2022-04-05 (Actual); Status verified 2022-03

CONDITIONS: Critical Illness; Near-Death Experience
MeSH Terms: conditions — Critical Illness; Death

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Greyson NDE scale — Questionnaire to detect occurence of NDE. A NDE is identified if score > or = 7/32
Diagnostic Test: DES dissociation scale — Screening for dissociative symptoms
Diagnostic Test: WHOQOL-SRPB — WHOQOL-SRPB is an instrument developed to evaluate how spirituality, religiosity and personal beliefs (SRPB) are related to quality of life in health and health care.
Diagnostic Test: cerebral magnetic resonance imaging — Types of images to be acquired: T1, T2, Diffusion Weighted Imaging-DWI, Fluid Attenuated Inversion Recovery and spectroscopy

SUMMARY:
This observational study aims to describe the incidence of near-death experience (NDE) in patients who survived a critical illness. In order to help determine the potential risk factors of NDE, dissociative status and spirituality are also investigated. Finally, in patients who experienced NDE, a magnetic resonance imaging is performed to search for any structural modifications.

ELIGIBILITY:
Inclusion Criteria:

* All consecutive patients who survived critical illness

Exclusion Criteria:

* Glasgow Coma Scale < 15/15
* Confusion (CAM ICU scale)
* Refusal

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All consecutive patients who survive any critical illness without exclusion criteria may be assessed for NDE occurence
Sampling Method: Non-Probability Sample
Enrollment: 126 (Actual)
Dates: Start 2019-06-01 (Actual); Primary Completion 2021-06-30 (Actual); Study Completion 2021-06-30 (Actual)

PRIMARY OUTCOMES:
NDE | Greyson questionnaire is administered during the week following ICU discharge
  NDE occurence during ICU stay, retrospectively detected by the Greyson scale. Greyson scale is a 16 items and 32 points scale. Minimal score is 0, maximal score is 32. A NDE is suspected when score is equal or higher than 7.

SECONDARY OUTCOMES:
Quality of life estimation | one year after first interview
  Quality of life assessment, using EQ-5D-3L
NDE | one year after first interview
  NDE occurence during ICU stay, retrospectively detected by the Greyson scale.
MCQ (Memory Characteristics Questionnaire) | one month after first interview
  analyze of the phenomenological characteristics of real and imagined memories

CONTACTS AND LOCATIONS:
Overall Officials: Anne-Françoise Rousseau, MD, PhD, Principal Investigator — University hospital of Liège
Locations (1):
- University Hospital of Liège, Liège, Belgium

REFERENCES:
- [Derived] Rousseau AF, Dams L, Massart Q, Choquer L, Cassol H, Laureys S, Misset B, Dardenne N, Gosseries O, Martial C. Incidence of near-death experiences in patients surviving a prolonged critical illness and their long-term impact: a prospective observational study. Crit Care. 2023 Feb 27;27(1):76. doi: 10.1186/s13054-023-04348-2. PMID 36849984